CLINICAL TRIAL: NCT07091227
Title: Efficacy and Safety of AK112 Combined Chemotherapy as Neoadjuvant Treatment for Signet Ring Cell-containing Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Efficacy and Safety of AK112 Combined Chemotherapy as Neoadjuvant Treatment for Signet Ring Cell-containing G/GEJ Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Akeso Biopharma Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K7937
Record Dates: First submitted 2025-07-02; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AK112+XELOX (Experimental): The participants received neoadjuvant therapy with AK112+oxaliplatin+capecitabine
  Interventions: Drug: AK112+oxaliplatin+capecitabine
- XELOX (Active Comparator): The participants received neoadjuvant therapy with oxaliplatin+capecitabine
  Interventions: Drug: oxaliplatin+capecitabine

INTERVENTIONS:
Drug: AK112+oxaliplatin+capecitabine — participants will receive standard dose treatment of AK112 combined with oxaliplatin+capecitabine every 3 weeks for 4 cycles before surgery.
  Other Names: AK112+XELOX
  Arms: AK112+XELOX
Drug: oxaliplatin+capecitabine — participants will receive standard dose treatment of oxaliplatin+capecitabine every 3 weeks for 4 cycles before surgery
  Other Names: XELOX
  Arms: XELOX

SUMMARY:
Study Overview

The primary objective of this clinical trial is to evaluate the efficacy and safety of AK112 in combination with chemotherapy as a neoadjuvant treatment for patients with locally advanced, resectable gastric or gastroesophageal junction (G/GEJ) adenocarcinoma containing signet ring cells.

Key Research Questions

1. Does neoadjuvant treatment with AK112 plus chemotherapy improve the pathological complete response (pCR) rate compared to chemotherapy alone in patients with locally advanced G/GEJ adenocarcinoma with signet ring cells?
2. What are the safety profile and additional efficacy outcomes of AK112 combined with chemotherapy in this patient population?

To answer these questions, the study will compare the combination of AK112 and chemotherapy with chemotherapy alone.

Participant Procedures

Eligible participants will:

1. Receive standard-dose AK112 in combination with chemotherapy every 3 weeks for a total of 4 cycles prior to surgery.
2. Undergo preoperative CT or MRI imaging within 3-4 weeks after the last treatment cycle to assess tumor response and evaluate eligibility for curative resection.
3. If no evidence of disease progression is observed and surgical evaluation is favorable, patients will undergo curative-intent gastrectomy within 6 weeks of completing neoadjuvant therapy (including oral agents, if any).
4. Postoperatively, adjuvant therapy will be administered at the investigator's discretion. Patients will be followed until disease recurrence or metastasis.
5. Attend clinic visits every 6 weeks during the neoadjuvant phase for evaluations and laboratory tests.
6. Maintain a symptom diary throughout the study period.
7. Undergo follow-up assessments every 3 months, starting from the first dose of study medication until 30 days after the last dose or the initiation of a new anti-tumor therapy.

Optional Imaging Substudy FAPI-PET/CT imaging will be explored as an optional diagnostic modality. Participation in this substudy will require separate informed consent and will be conducted under a future protocol amendment (pending IRB approval).

ELIGIBILITY:
Inclusion Criteria

1. Subjects must voluntarily agree to participate in the clinical trial and sign a written informed consent form (ICF) before undergoing any trial-related procedures.
2. Male or female subjects aged ≥18 and ≤75 years at the time of signing the informed consent.
3. Histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction with signet ring cell components. Diagnosis of locally advanced disease (based on AJCC 8th edition) must be made within 4 weeks prior to randomization.
4. Tumor staging: cT3-4a or cN+ (M0) as determined by endoscopic ultrasound and/or contrast-enhanced CT/MRI. Diagnostic laparoscopy may be used as needed. The tumor must be assessed as resectable by the investigator.
5. Immunohistochemical testing confirms proficient mismatch repair (pMMR) status and HER-2 negativity (IHC 0 or 1+, or IHC 2+ with negative FISH for HER-2 amplification).
6. No prior systemic treatment for the current malignancy, including surgery, chemotherapy, radiotherapy, or immunotherapy.
7. Eligible for radical surgery with no surgical contraindications as determined by a qualified surgeon.
8. ECOG performance status of 0 or 1 within 7 days before randomization.
9. Estimated life expectancy > 6 months.
10. Adequate organ function, as demonstrated by the following laboratory results (without blood product transfusion or cytokine support within 2 weeks prior to first dose):

Hematologic: WBC ≥ 3.5 × 10⁹/L, ANC ≥ 1.5 × 10⁹/L, Platelets ≥ 100 × 10⁹/L, Hemoglobin ≥ 90 g/L Hepatic: Total bilirubin ≤ 1.5 × ULN, AST and ALT ≤ 2.5 × ULN Renal: Serum creatinine ≤ 1.0 × ULN, Creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula) Coagulation: INR, APTT, PT ≤ 1.5 × ULN Thyroid: TSH within normal limits. If TSH is abnormal, subjects with normal total T3 (or FT3) and FT4 may be enrolled.

Cardiac: Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram; cardiac assessment may be required for patients with cardiac comorbidities.

Hepatitis B serology: HBsAg (-) and anti-HBc (-). If HBsAg (+) or anti-HBc (+), HBV-DNA must be <1000 copies/mL or <200 IU/mL or below the site-specific ULN.

HCV antibody (-). Subjects with positive HCV antibody but negative HCV-RNA may be considered eligible.

11) For women of childbearing potential: Negative serum or urine pregnancy test within 7 days before randomization. If urine test is inconclusive, a serum test is required. Postmenopausal status is defined as ≥12 months of amenorrhea or surgical sterilization (bilateral oophorectomy/hysterectomy).

12) Subjects (regardless of sex) with reproductive potential must agree to use highly effective contraception (failure rate <1%) from the start of study treatment to 120 days after last study dose (or 180 days if receiving chemotherapy).

13) Breastfeeding is not permitted during the study period.

Exclusion Criteria

1. Histology other than adenocarcinoma with signet ring cell features, including squamous cell carcinoma, neuroendocrine carcinoma, or other subtypes.
2. Tumor exhibiting deficient MMR (dMMR) or HER-2 positivity (IHC 3+, or IHC 2+ with FISH-confirmed HER-2 amplification).
3. Unresectable tumors or subjects unwilling or unable to undergo surgery due to medical, anatomical, or personal reasons.
4. History of other malignancies within 5 years prior to enrollment, excluding certain cured cancers (e.g., basal cell carcinoma, carcinoma in situ of cervix/breast/prostate/bladder).
5. Evidence of active bleeding on endoscopy.
6. Participation in another interventional clinical study or use of investigational drugs/devices within 4 weeks prior to enrollment.
7. Prior immunotherapy including immune checkpoint inhibitors (e.g., anti-PD-1/PD-L1, anti-CTLA-4, anti-TIGIT, etc.) or cellular immunotherapy.
8. Use of traditional Chinese medicine with antitumor or immunomodulatory effects within 2 weeks prior to first dose.
9. Active autoimmune disease requiring systemic therapy in the last 2 years. Hormonal replacement therapies are allowed.
10. Use of systemic corticosteroids or immunosuppressants within 7 days before first dose (except ≤10 mg/day prednisone equivalent).
11. Prior or planned organ/bone marrow transplantation (excluding corneal transplant).
12. Known hypersensitivity to investigational products.
13. Conditions affecting oral administration of capecitabine (e.g., dysphagia, intestinal obstruction).
14. HIV infection (HIV-1/2 antibody positive).
15. Active hepatitis B (HBsAg positive and HBV DNA > ULN).
16. Active hepatitis C (HCV antibody positive with detectable HCV RNA).
17. Receipt of live vaccines within 30 days prior to first dose. Inactivated influenza vaccines are permitted; live attenuated intranasal influenza vaccine is not.
18. Pregnant or breastfeeding women.
19. Serious or uncontrolled systemic illnesses, including:

    Significant arrhythmias or heart block

    History of myocarditis, cardiomyopathy, MI, unstable angina, CHF within 12 months

    Gastrointestinal conditions (e.g., active ulcers, varices, perforation, abscess) within 6 months

    Recent COPD exacerbation (within 1 month)

    Grade ≥3 thromboembolic events or cerebrovascular accidents within 6 months

    Poorly controlled hypertension (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg despite treatment)

    Non-infectious pneumonitis or interstitial lung disease

    Pulmonary tuberculosis

    Active systemic infection

    Decompensated liver disease

    Poorly controlled diabetes (FBG >10 mmol/L or random BG >16 mmol/L)

    Proteinuria ≥ ++ or 24-hour urine protein > 1.0 g
20. Psychiatric illness interfering with compliance or safety.
21. Major surgery or significant trauma within 30 days prior to first dose, or planned major surgery within 30 days post first dose (except minor procedures).
22. Tumor necrosis on imaging, deemed high risk for bleeding by investigator.
23. History of severe bleeding or coagulation disorders; active bleeding within 1 month (e.g., hematemesis, hemoptysis, significant epistaxis); long-term anticoagulation for atrial fibrillation with CHADS2 ≥ 2.
24. Any condition or laboratory abnormality that, in the opinion of the investigator, may interfere with the study results or subject safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-07-20 (Estimated); Study Completion 2029-07-20 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | At surgery
  Absence of viable tumor cells in primary tumor and lymph nodes (Becker TRG 1a)

SECONDARY OUTCOMES:
Objective Response Rate，ORR | After 2 neoadjuvant cycles (6 weeks), and 4 neoadjuvant cycles(12 weeks)
  Proportion of participants achieving CR or PR per RECIST v1.1 assessed via contrast-enhanced CT/MRI
Disease-Free Survival, DFS | Assessed every 12 weeks via CT/MRI up to 60 months from postoperative.
  The time between postoperative and disease recurrence or (for any reason) death.
Treatment-Emergent Adverse Events (TEAEs) | First dose to 90 days post-surgery
  Incidence of adverse events graded by CTCAE v6.0
Serious Adverse Events (SAE) | First dose to 90 days post-surgery
  Serious AEs leading to discontinuation
R0 Resection Rate | At surgery
  Percentage of participants achieving microscopically margin-negative resection

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, Principal Investigator — Department of Cancer Medical Center, Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing，100730
Locations (1):
- Department of Cancer Medical Center, Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying published results (including baseline characteristics, outcome measures, and protocol deviations) will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after primary publication and available for 10 years
Access Criteria: 1. Researchers must submit a methodologically sound proposal to [DataAccess@PUMCH.cn](mailto:DataAccess@PUMCH.cn)
  2. Approval by the sponsor's independent data access committee
  3. Signed data sharing agreement
  4. Proposals may be rejected for commercial/competitive reasons
URL: http://DataAccess@PUMCH.cn